CLINICAL TRIAL: NCT05584254
Title: Effects of β-glucan Based Dietary Fibres on Indomethacin-induced Hyperpermeability and Gut Microbiota Composition in Elderly: A Randomized Placebo-controlled Crossover Clinical Trial
Brief Title: Effects of β-glucans on Gut Permeability and Microbiota in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Kerry Group (Unknown)
Responsible Party: Principal Investigator, Robert Brummer, Professor, MD, Örebro University, Sweden
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FODI
Record Dates: First submitted 2022-10-03; First posted 2022-10-18 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Elderly; Bowel Symptoms; Prebiotics
Keywords: elderly; prebiotics; permeability; clinical trial; Microbiota; Health

STUDY DESIGN:
Intervention Model Description: 3 study products (2 different forms of yeast-beta glucan and a placebo) taken in a cross-over design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elderly with gastrointestinal symptoms (Experimental): The target group for the intervention and cohort of interest used for comparison of baseline characteristics between control groups. Went into a cross-over design with 2 yeast-derived beta-glucan supplements and a placebo.
  Interventions: Dietary Supplement: yeast-beta glucan
- Senior orienteers (No Intervention): A model of healthy aged elderly used as a control group for the baseline characteristics.
- Young healthy adults (No Intervention): A cohort of young healthy adults used as a control group for the baseline characteristics.

INTERVENTIONS:
Dietary Supplement: yeast-beta glucan
  Arms: Elderly with gastrointestinal symptoms

SUMMARY:
The investigators aim was to compare healthy young adults, senior orienteers (model of healthy ageing) and elderly with gastrointestinal symptoms on intestinal permeability, microbiota compositions and well-being. In addition, assess whether 3 weeks of oral intake of soluble or dispersible forms yeast-dervied beta-glucan could improve intestinal barrier function against drug-induced barrier disruption vs placebo for a cohort of elderly people with gastrointestinal symptoms, in a randomized double blinded placebo-controlled cross-over clinical trial.

DETAILED DESCRIPTION:
Baseline samples for measurements of intestinal permeability (multisugar test), microbiota composition (faecal samples) and well-being (questionnaires) were collected during the first week for:

Young healthy adults (healthy young controls) Senior orienteers (healthy elderly controls) Elderly with gastrointestinal (GI) symptoms

Thereafter only the elderly with GI symptoms continued into the randomized cross-over trial where they were blindly and randomly distributed one of the following: Soluble yeast-derived beta-glucan, dispersible (whole) yeast-derived beta-glucan and placebo. Each supplement was taken for 3 weeks with a 1 week washout until all participants had taken all supplements. Towards the end of each supplement period, samples for measurement of intestinal permeability and microbiota were collected, in addition to questionnaires being filled out.

ELIGIBILITY:
Elderly with gastrointestinal symptoms

Inclusion Criteria:

* Informed consent signed by study participant
* Age >55 years
* Scoring above 2 on the dimensions for diarrhoea and constipation on the Gastrointestinal symptoms rating scale (GSRS)
* Mentally and physically fit to complete questionnaires during the study period

Exclusion Criteria:

* Known or genic gastrointestinal diseasewith strictures, malignance's and ischemia.
* Inflammatory bowel diseases (IBD)
* Participation in other clinical trials in the past three months.
* Intake of medications know to change the inflammatory status (i.e proton pump inhibitors, antibiotic, anti-inflammtory medication (including NSAIDs)

Healthy controls

Inclusion Criteria:

* Age ≥ 18 years
* Informed consent signed by the study participant
* Mentally and physically fit to complete questionnaires during the study period

Exclusion Criteria:

* Previous abdominal surgery
* A hypertonic condition demanding medical treatment
* Diagnosed psychiatric disease
* Lactose intolerance
* Usage of medical prescribed medications, expect oral contraceptives, during the 14 days preceding study start
* Premenstrual syndrome
* Pregnant or breast feeding
* Known or genic gastrointestinal disease, with strictures, malignance's and ischemia.
* Inflammatory bowel diseases (IBD)
* Participation in other clinical trials in the past three months.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability at baseline (before indomethacin) | Day 1
  In vivo gastrointestinal permeability measured by oral intake of multi-sugar test before intake of indomethacin. Urine collected over 24 hours for measurement of excreted sugars.
Intestinal permeability at baseline (after indomethacin) | Day 1
  In vivo gastrointestinal (GI) permeability measured by oral intake of multi-sugar test after intake of indomethacin (GI barrier disruption challenge). Urine collected over 24 hours for measurement of excreted sugars.
Changes in Intestinal permeability 3 weeks after study supplementation 1 (before indomethacin). | 3 weeks
  Performed after study participants have orally taken study supplementation 1 for 3 weeks. In vivo gastrointestinal permeability measured by oral intake of multi-sugar test before intake of indomethacin. Urine collected over 24 hours for measurement of excreted sugars.
Changes in intestinal permeability 3 weeks after study supplementation 1 (after indomethacin). | 3 weeks
  Performed after study participants have orally taken study supplementation 1 for 3 weeks.
  In vivo gastrointestinal (GI) permeability measured by oral intake of multi-sugar test after intake of indomethacin (GI barrier disruption challenge). Urine collected over 24 hours for measurement of excreted sugars.
Changes in intestinal permeability 3 weeks after study supplementation 2 (before indomethacin) | 3 weeks
  Performed after study participants have orally taken study supplementation 2 for 3 weeks.
  In vivo gastrointestinal permeability measured by oral intake of multi-sugar test before intake of indomethacin. Urine collected over 24 hours for measurement of excreted sugars.
Changes in intestinal permeability 3 weeks after study supplementation 2 (after indomethacin) | 3 weeks
  Performed after study participants have orally taken study supplementation 2 for 3 weeks.
  In vivo gastrointestinal (GI) permeability measured by oral intake of multi-sugar test after intake of indomethacin (GI barrier disruption challenge). Urine collected over 24 hours for measurement of excreted sugars.
Changes in intestinal permeability 3 weeks after study supplementation 3 (before indomethacin) | 3 weeks
  Performed after study participants have orally taken study supplementation 3 for 3 weeks.
  In vivo gastrointestinal permeability measured by oral intake of multi-sugar test before intake of indomethacin. Urine collected over 24 hours for measurement of excreted sugars.
Changes in intestinal permeability 3 weeks after study supplementation 3 (after indomethacin) | 3 weeks
  Performed after study participants have orally taken study supplementation 3 for 3 weeks.
  In vivo gastrointestinal (GI) permeability measured by oral intake of multi-sugar test after intake of indomethacin (GI barrier disruption challenge). Urine collected over 24 hours for measurement of excreted sugars.

SECONDARY OUTCOMES:
Microbiota diversity - at baseline | Day 1
  Faecal samples will be used for next-generation sequencing and analysed for diversity
Bacterial species - at baseline | Day 1
  Faecal samples will be used for next-generation sequencing and analysed for bacterial species
Changes in microbiota diversity 3 weeks after study supplementation 1 | 3 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in microbiota diversity
Changes in bacterial species 3 weeks after study supplementation 1 | 3 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in bacterial species levels
Changes in microbiota diversity 3 weeks after study supplementation 2 | 3 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in microbiota diversity
Changes in bacterial species 3 weeks after study supplementation 2 | 3 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in bacterial species levels
Changes in microbiota diversity 3 weeks after study supplementation 3 | 3 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in microbiota diversity
Changes in bacterial species 3 weeks after study supplementation 3 | 3 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in bacterial species levels
Changes in microbiota diversity - Washout (1 week after ending supplementation 1, i.e. 4 weeks after baseline) | 4 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in microbiota diversity from 1 weeks washout, after ending study supplementation 1 (4 weeks after baseline)
Changes in bacterial species - Washout (1 week after ending study supplementation 1, i.e. 4 weeks after baseline) | 4 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in bacterial species from 1 weeks washout, after ending study supplementation 1 (4 weeks after baseline)
Changes in microbiota diversity - Washout (1 week after ending study supplementation 2, i.e. 4 weeks after baseline) | 4 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in microbiota diversity from 1 weeks washout, after ending study supplementation 2 (4 weeks after baseline)
Changes in bacterial species - Washout (1 week after ending study supplementation 2, i.e. 4 weeks after baseline) | 4 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in bacterial species from 1 weeks washout, after ending study supplementation 2 (4 weeks after baseline).
Changes in microbiota diversity - Washout (1 week after ending study supplementation 3, i.e. 4 weeks after baseline) | 4 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in microbiota diversity from 1 weeks washout, after ending study supplementation 3 (4 weeks after baseline)
Changes in bacterial species - Washout (1 week after ending study supplementation 3, i.e. 4 weeks after baseline) | 4 weeks
  Faecal samples will be used for next-generation sequencing and analysed for changes in bacterial species from 1 weeks washout, after ending study supplementation 3 (4 weeks after baseline)
Changes in gastrointestinal symptom questionnaire scores | up to 13 weeks
  The Gastrointestinal Symptoms Rating Scale (GSRS) evaluates gastrointestinal (GI) symptoms based on the 5 domains diarrhoea, constipation, reflux, indigestion and abdominal pain. The symptoms are assessed with 15 items, ranging in scores 1 to 7 depending on their severity. A score of 1 represents "no problems" and score 7 represents "severe problems". The severity of symptoms may be defined as no problems (1 point), mild (1-2 points), moderate (2-4 points), and severe (4-7 points). The scores for each domain was calculated as the mean score of each corresponding item while the mean total GSRS score reflects the general severity of GI symptoms.
Changes in hospital and anxiety depression scores | up to 13 weeks
  The Hospital Anxiety and Depression Scale (HADS) was used to evaluate the psychological distress of study participants.This questionnaire consists of 14 items subdivided in two subscales for the assessment of anxiety or depression. The total score is used as a measure of general psychological distress. The minimum score is 0 and the maximum score is 21. A score > 8 on respective subscales indicates a significant level of anxiety or depression.
Changes in perceived stress scale scores | Up to 13 weeks
  The perceived stress scale (PSS) consists of 10 items, including a number of direct questions about current levels of experienced stress. The respondent answers how often a certain emotion has been present during the past month. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Each item is rated on a 5-point scale ranging from never (0) to almost always (4). The questions in this scale ask about the responders feelings and thoughts during the last month. In each case the questionnaire requires the respondent to indicate by circling how often they felt or thought a certain way.
Changes in quality of life questionnaire scores | Up to 13 weeks
  The EuroQol 5D-5L (EQ-5D-5L) tool consists of two parts; 5Q-5D, which includes 5 items related to wellbeing and function (mobility, self-care, usual activities, pain/discomfort and anxiety/ depression) and the visual analogue scale, 5Q-5D-VAS, ranging from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, PhD/MD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Campus USÖ, Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No